CLINICAL TRIAL: NCT01555762
Title: Non Interventional Study Evaluating Efficacy and Safety in a Cohort of Elderly Patients of First Line Therapy With Avastin ® Regimen for Metastatic Colorectal Cancer.
Brief Title: An Observational Study of Avastin in First Line in Elderly Patients With Metastatic Colorectal Cancer (CASSIOPEE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27829
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, prospective, observational study will evaluate the efficacy and safety of Avastin (bevacizumab) in first-line therapy in elderly patients with metastatic colorectal cancer. Data will be collected from eligible patients for24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 75 years of age
* Metastatic colorectal cancer
* Initiating Avastin first-line therapy in combination with chemotherapy

Exclusion Criteria:

* Previous Avastin therapy
* Patient participating in a clinical study evaluating a cytotoxic anti-cancer therapy and/or an investigational new drug

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with metastatic colorectal cancer initiating first-line treatment with Avastin
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (166):
- France (166):
  - Ch D Abbeville; Medecine B1, Abbeville
  - Clinique Du Docteur Calabet; Cromg, Agen
  - Ch D Agen; Medecine Interne II, Agen
  - C.H. Du Pays D'aix En Provence Service du Dr Blanc, Aix-en-Provence
  - Poly Parc Rambot La Provencale; Chimiotherapie Ambulatoire, Aix-en-Provence
  - Chd Castelluccio; Oncologie, Ajaccio
  - Clinique Claude Bernard; Onco Hematologie, Albi
  - Chi D Alencon; Medecine Ambulatoire, Alençon
  - Chi D Alencon; Medecine I, Alençon
  - Hopital Nord; Medecine A, Amiens
  - Clinique De L Europe; Pmsi, Amiens
  - Clinique De L Europe; Radiotherapie Chimiotherapie, Amiens
  - Centre Hospitalier de L'Agglomeration Montargeoise; Medecine Polyvalente A Orientation Mi & Cancero, Amilly
  - Cham; Medecine D, Amilly
  - Ctre Radiotherapie Et Onco Medic, Amilly
  - Hotel Dieu; Medecine A, Angers
  - Cabinet Medical, Arras
  - Centre Radiotherapie Marie Curie, Arras
  - Ch D Ardeche Meridionale; Medecine A2, Aubenas
  - Ch D Auch; Med Interne Chimiotherapie, Auch
  - Clinique Sainte Catherine; Hopital De Semaine, Avignon
  - Clinique Du Docteur Maymard; Hopital De Jour Chimiotherapie, Bastia
  - Hopital De Falconaja Furiani; Hopital De Jour, Bastia
  - Centre Hospitalier de La Cote Basque; Oncologie, Bayonne
  - Centre Hospitalier; Hematologie-Oncologie, Beauvais
  - Hopital Jean Minjoz; Gastro Enterologie, Besançon
  - Hopital Jean Minjoz; Hopital de Jour, Besançon
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Clinique Anne D Artois; Gastro Enterologie, Béthune
  - Clinique Champeau Mediterranee; Radiotherapie Oncologie, Béziers
  - Hopital Avicenne; Cancerologie, Bobigny
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Polyclin Bordeaux Nord Aquitaine; Gastro Enterologie, Bordeaux
  - Centre Hospitalier Dr Duchenne; Hepato Gastro Enterologie, Boulogne-sur-Mer
  - Clinique Du Docteur Convert; Medecine, Bourg-en-Bresse
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Ch De Fleyriat; Gastro Enterologie, Bourg-en-Bresse
  - Hopital Augustin Morvan; Federation De Cancerologie, Brest
  - Clinique Pasteur Lanroze; Chimiotherapie Radiotherapie, Brest
  - CMC de Bligny; Hopital de Jour, Briis-sous-Forges
  - CMC de Bligny; Oncologie Court Sejour, Briis-sous-Forges
  - CMC de Bligny; Oncologie SSR, Briis-sous-Forges
  - Ch De Brive La Gaillarde; Radiotherapie Oncologie, Brive-la-Gaillarde
  - Hopital Cote De Nacre; Gastro Enterologie, Caen
  - Infirmerie Protestante; Endos Digestive Coelioscopie, Caluire-et-Cuire
  - Hopital Pierre Nouveau; Medecine A, Cannes
  - Ch Antoine Gayraud; Oncologie, Carcassonne
  - Clinique Montreal; Chimiotherapie, Carcassonne
  - Clinique Du Parc; Hematologie, Castelnau Lez
  - Cabinet Medical, Challes-les-Eaux
  - Medipole De Savoie; Departement Oncologie, Challes-les-Eaux
  - Oncologie 37; Bureau, Chambray-lès-Tours
  - Hopital Prive Paul d Egine; Chimiotherapie Ambulatoire, Champigny-sur-Marne
  - Centre Hospitalier; Oncologie, Châteauroux
  - Ch De Cholet; Gastro Enterologie, Cholet
  - Pole Sante Republique;Oncologie Hematologie, Clermont-Ferrand
  - Hopital Louis Pasteur; Medecine A, Colmar
  - Polyclinique Saint Come; Hopital De Jour Oncologie, Compiègne
  - CH Sud Francilien; Oncologie, Corbeil-Essonnes
  - Ch Laennec; Medecine V, Creil
  - CHU Henri Mondor; Service d'Oncologie Medicale, Créteil
  - Ch De Dax; Radiotherapie Oncologie, Dax
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Hopital Victor Jousselin; Gastro Enterologie, Druex
  - Centre D Oncologie Dunkerquois, Dunkirk
  - Chi Eure Seine D Evreux; Oncologie Conventionnelle, Évreux
  - Clinique Pasteur; Oncologie Medicale, Hematologie, Évreux
  - Ch Jacques Monod;Medecine A4 B4, Flers
  - Hopital De Freyming; Secteur 1, Freyming-Merlebach
  - Chi De Frejus Saint Raphael; Hopital De Jour, Fréjus
  - Chi Alpes Du Sud Site De Gap; Med Interne Et Polyvalente, Gap
  - Centre Gastro Loire, Gien
  - Hopital Nord Ouest;Gastro Enterologie, Gleizé
  - CH Emmanuel Rain; Oncologie, Gonesse
  - Hopital Prive De Chantilly; Medecine, Gouvieux Chantilly
  - Hopital Alpha Sante De Hayange; Medecine B, Hayange
  - Clinique Sainte Marguerite; Oncologie Medicale, Hyères
  - Polyclinique de Blois; Chimiotherapie Ambulatoire, La Chaussée-Saint-Victor
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Saint Louis; Oncologie Medicale, La Rochelle
  - Hopital Albert Michallon; Oncologie, La Tronche
  - Hopital Albert Michallon; Radiotherapie, La Tronche
  - Ch De Lagny Sur Marne; Oncologie, Lagny-sur-Marne
  - Hopital Robert Boulin; Oncologie, Libourne
  - Polyclinique Du Bois; Oncologie, Lille
  - Polyclinique De La Louviere; Chimiotherapie, Lille
  - Ch De Longjumeau; Hopital De Jour Et Semaine, Longjumeau
  - Clinique Des 4 Pavillons; Chimiotherapie, Lormont
  - Hopital De La Croix Rousse;Hepato Gastro Entero, Lyon
  - Ctre Consultations La Sauvegarde, Lyon
  - Ctre Hosp St Joseph Et St Luc; Gastro Enterologie Endoscopie, Lyon
  - Hopital Prive Jean Mermoz; Cancerologie, Lyon
  - Hopital Prive Jean Mermoz; Gastro Enterologie Hepatologie, Lyon
  - Clin Mut De Lyon Eugene Andre; Hopital De Jour 1er B, Lyon
  - Hopital Edouard Herriot; Pavillon E Oncologie Medicale, Lyon
  - Clinique Saint Francois; Oncologie Medicale, Mainvilliers
  - Clinique Mutualiste Bonneveine; Oncologie Medicale, Marseille
  - CH Prive Clairval; Chimiotherapie Ambulatoire, Marseille
  - Hôpital Saint Joseph; Oncologie Medicale, Marseille
  - Hopital Timone Adultes; Oncologie Digestive, Marseille
  - Clinique Du Parc; Centre de Radiotherapie Gray, Maubeuge
  - Hopital Clinique Claude Bernard; Oncologie Medicale, Metz
  - Chra; Gastro Enterologie, Metz-Tessy
  - Hopital Layne; Medecine A2, Mont-de-Marsan
  - Hopital Layne; Medecine Ambulatoire, Mont-de-Marsan
  - Ch De Montauban; Medecine Interne, Montauban
  - Site Le Mittan; Hopital De Jour, Montbéliard
  - Ch De Montelimar; Gastro Enterologie Oncologie, Montélimar
  - Ghi Le Raincy Montfermeil; Gastro Medecine Interne, Montfermeil
  - Ghi Le Raincy Montfermeil; Radiotherapie Oncologie, Montfermeil
  - Hopital Jacques Monod; Hopital De Semaine Unite 53, Montivilliers
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Hopital Saint Eloi; Hopital De Jour, Montpellier
  - Polyclinique Saint Roch; Hop Jour Chimio Radiotherapie, Montpellier
  - Centre Azureen De Cancerologie; Cons externes, Mougins
  - Clinique D Occitanie; Chimiotherapie Ambulatoire, Muret
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Polyclinique Du Languedoc; Chimiotherapie, Narbonne
  - Hopital Americain; Sce Oncologie, Neuilly-sur-Seine
  - Ctre Radiotherapie Cyr Deguergue, Nevers
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Hopital Caremeau; Gastro Enterologie, Nîmes
  - Hopital Prive Armand Brillard; Groupe Sein Paris Est, Nogent-sur-Marne
  - Polyclinique Des Murlins;Ambulatoire, Orléans
  - Clinique sainte marie; chimiotherapie ambulatoire, Osny
  - Hopital Des Diaconesses; Oncologie, Paris
  - Hopital Saint Antoine; Oncologie Medicale, Paris
  - CH Pitie Salpetriere; Hepathologie Gastro Enterologie, Paris
  - GH Paris Saint Joseph; Hopital De Jour Oncologie, Paris
  - Hopital Bichat Claude Bernard; Hepatologie Gastro Enterologie, Paris
  - Hop Europeen Georges Pompidou; Gastro Enterologie, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Hopital Saint Jean; Hospitalisation Oncologie, Perpignan
  - Hopital Du Haut-Leveque; Gastro-Enterologie, Pessac
  - Clinique Francheville; Radiotherapie, Périgueux
  - Polyclinique Francheville; MED CHIMIOTHERAPIE RADIOTHERAPIE, Périgueux
  - Ch Lyon Sud; Chir Visc Sect Jules Courmont, Pierre-Bénite
  - Ch Lyon Sud; Gastro Secteur Jules Courmont, Pierre-Bénite
  - Ctre Hosp Des Vals D Ardeche; Medecine C, Privas
  - Ch De Rambouillet; Medecine A2, Rambouillet
  - Ch Arrondissement De Montreuil; Medecine 1, Rang-du-Fliers
  - Centre Frederic Joliot Curie, Rouen
  - Hopital Yves Le Foll; Hematologie Oncologie, Saint-Brieuc
  - Ctre De Radiotherapie St Vincent, Saint-Grégoire
  - Clinique de L'Union; Oncologie, Saint-Jean
  - Memorial France Etats Unis; Hopital De Jour, Saint-Lô
  - Centre Joliot Curie, Saint-Martin-Boulogne
  - Ch De Saint Quentin; Gastro Enterologie Endoscopie, Saint-Quentin
  - Ch De Selestat; Medecine A, Sélestat
  - Centre Clinical; Oncologie Medicale, Soyaux
  - Hopital Broussais; Medecine 2A, St-Malo
  - Clinique Chir De L Orangerie; Chimiotherapie, Strasbourg
  - Clinique Saint Anne; Hopital De Jour, Strasbourg
  - Fondation Maison Sante Bagatelle; Gastro Enterologie, Talence
  - Hopitaux Du Leman Site Thonon; Gastro Enterologie, Thonon-les-Bains
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Hopital Joseph Ducuing; Medecine Interne, Toulouse
  - Hopital Prive Du Vert Galant; Cons Specialisees, Tremblay-en-France
  - Ch De Valence; Medecine 6, Valence
  - Clinique Oceane; Medecine B, Vannes
  - Hopital Saint Nicolas; Medecine A, Verdun
  - Clinique De La Porte Verte; EST 3, Versailles
  - Gh Mutualiste Les Portes Du Sud; Gastro-Enterologie, Vénissieux
  - Hopital Prive Villeneuve d Ascq;Chimiotherapie Radiotherapie, Villeneuve-d'Ascq

REFERENCES:
- [Derived] Francois E, Mineur L, Deplanque G, Laplaige P, Smith D, Gourgou S, Tanang A, Ionescu-Goga M, Veerabudun K, Lelarge Y, Kim S, Rollot F. Efficacy and Safety of Bevacizumab Combined With First-Line Chemotherapy in Elderly (>/=75 Years) Patients With Metastatic Colorectal Cancer: A Real-World Study. Clin Colorectal Cancer. 2020 Sep;19(3):e100-e109. doi: 10.1016/j.clcc.2020.02.009. Epub 2020 Apr 13. PMID 32299778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 402 participants were enrolled from 100 French sites.
Pre-assignment Details: The data in the study for participant flow, baseline characteristics, outcome measure and adverse events was collected for overall participants and not as per the dose administered to participants.
Groups:
- Bevacizumab: Participants received initial dose of either 5 milligram per kilogram (mg/kg) every 2 weeks or 7.5 mg/kg every 3 weeks of bevacizumab irrespective of the age subgroup.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 402
Safety Population | 383
Efficacy Population | 358
Completed | 128
Not Completed | 274
Not completed — No information on Bevacizumab intake | 11
Not completed — Missing start date of infusion | 8
Not completed — 75 years old or more ticked No | 1
Not completed — Treatment with Bevacizumab ticked No | 24
Not completed — Death linked to progression of disease | 165
Not completed — Lost follow-up/moved house/changed team | 35
Not completed — Investigator's decision | 10
Not completed — Participant not wishing to continue | 5
Not completed — Missing data | 1
Not completed — Death linked to an adverse event | 14

BASELINE CHARACTERISTICS:
Population: The efficacy population included all participants who had at least one infusion of bevacizumab, without exclusion criteria and excluding participants with no intake of chemotherapy, or intake of bevacizumab before or 2 months after chemotherapy initiation. Data in the study was collected for overall participants and not as per dose administered.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.5 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 185

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the time of first dose of study treatment to the time of disease progression or death from any cause (Up to 53 months)
Population: The efficacy population (EFF) included all participants who had at least one infusion of bevacizumab, without exclusion criteria and excluding participants with no intake of chemotherapy, or intake of bevacizumab before or 2 months after chemotherapy initiation. Data in study was collected for overall participants and not as per dose administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
Months | 9.14 [8.32 to 10.16]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time between the treatment start date (date of the first infusion of bevacizumab) and date of all-cause death.
Time Frame: From the time of first dose of study treatment to the time of death from any cause (Up to 53 months)
Population: The EFF included all participants who had at least one infusion of bevacizumab, without exclusion criteria and excluding participants with no intake of chemotherapy, or intake of bevacizumab before or 2 months after chemotherapy initiation. Data in the study was collected for overall participants and not as per dose administered to participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
Months | 19.00 [16.47 to 21.47]

3. Secondary Outcome: Percentage of Participants With Bevacizumab Administration
Time Frame: Up to 36 months
Population: The EFF included all participants who had at least one infusion of bevacizumab, without exclusion criteria and excluding participants with no intake of chemotherapy, or intake of bevacizumab before or 2 months after chemotherapy initiation.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
Percentage of participants
  5 mg/kg/2 weeks: number analyzed (Participants) | 357
  5 mg/kg/2 weeks | 90.8
  7.5 mg/kg/3 weeks: number analyzed (Participants) | 357
  7.5 mg/kg/3 weeks | 7.3
  At least one change in dosing | 1.7
  At least one temporary discontinuation | 12.3
  Permanent discontinuation | 82.4

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: Up to 53 months
Population: Safety population included all participants who had at least one infusion of bevacizumab. Data in the study was collected for overall participants and not as per dose administered to participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 383
Percentage of participants | 60.8

5. Secondary Outcome: Percentage of Participants With Activities of Daily Living (ADL)
Description: The Katz Activity of Daily Living (ADL) questionnaire scale contains 6 items evaluating in terms of autonomy or dependence the patient's ability to carry out basic activities of daily living (bathing, dressing, toileting, transfer, continence, feeding). Total score range 0 (low) to 6 (high). High score indicates participant is independent.
Time Frame: Baseline, Month 6, 12, 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
Percentage of participants
  Baseline: Bathing (self-sufficient): number analyzed (Participants) | 353
  Baseline: Bathing (self-sufficient) | 89.2
  Baseline: Bathing (partial help): number analyzed (Participants) | 353
  Baseline: Bathing (partial help) | 8.2
  Baseline: Bathing (washing impossible): number analyzed (Participants) | 353
  Baseline: Bathing (washing impossible) | 2.5
  Baseline: Dressing (self-sufficient): number analyzed (Participants) | 354
  Baseline: Dressing (self-sufficient) | 92.9
  Baseline: Dressing (partial help): number analyzed (Participants) | 354
  Baseline: Dressing (partial help) | 4.2
  Baseline: Dressing (completely undressed): number analyzed (Participants) | 354
  Baseline: Dressing (completely undressed) | 2.8
  Baseline: Toileting (self-sufficient): number analyzed (Participants) | 354
  Baseline: Toileting (self-sufficient) | 95.8
  Baseline: Toileting (needs help): number analyzed (Participants) | 354
  Baseline: Toileting (needs help) | 2.5
  Baseline: Toileting (doesn't go): number analyzed (Participants) | 354
  Baseline: Toileting (doesn't go) | 1.7
  Baseline: Transfer (self-sufficient): number analyzed (Participants) | 354
  Baseline: Transfer (self-sufficient) | 90.7
  Baseline: Transfer (needs help): number analyzed (Participants) | 354
  Baseline: Transfer (needs help) | 8.2
  Baseline: Transfer (bedridden): number analyzed (Participants) | 354
  Baseline: Transfer (bedridden) | 1.1
  Baseline: Cont (continent): number analyzed (Participants) | 351
  Baseline: Cont (continent) | 86.6
  Baseline:Cont (occasional incontinence): number analyzed (Participants) | 351
  Baseline:Cont (occasional incontinence) | 12.3
  Baseline:Cont (permanent incontinence): number analyzed (Participants) | 351
  Baseline:Cont (permanent incontinence) | 1.1
  Baseline: Feeding (self-sufficient): number analyzed (Participants) | 354
  Baseline: Feeding (self-sufficient) | 96.6
  Baseline: Feeding (needs help): number analyzed (Participants) | 354
  Baseline: Feeding (needs help) | 3.4
  Month 6: Bathing (self-sufficient): number analyzed (Participants) | 260
  Month 6: Bathing (self-sufficient) | 85.4
  Month 6: Bathing (partial help): number analyzed (Participants) | 260
  Month 6: Bathing (partial help) | 13.1
  Month 6: Bathing (washing impossible): number analyzed (Participants) | 260
  Month 6: Bathing (washing impossible) | 1.5
  Month 6: Dressing (self-sufficient): number analyzed (Participants) | 260
  Month 6: Dressing (self-sufficient) | 91.9
  Month 6: Dressing (partial help): number analyzed (Participants) | 260
  Month 6: Dressing (partial help) | 6.5
  Month 6: Dressing (completely undressed): number analyzed (Participants) | 260
  Month 6: Dressing (completely undressed) | 1.5
  Month 6: Toileting (self-sufficient): number analyzed (Participants) | 260
  Month 6: Toileting (self-sufficient) | 95.0
  Month 6: Toileting (needs help): number analyzed (Participants) | 260
  Month 6: Toileting (needs help) | 4.6
  Month 6: Toileting (doesn't go): number analyzed (Participants) | 260
  Month 6: Toileting (doesn't go) | 0.4
  Month 6: Transfer (self-sufficient): number analyzed (Participants) | 260
  Month 6: Transfer (self-sufficient) | 91.2
  Month 6: Transfer (needs help): number analyzed (Participants) | 260
  Month 6: Transfer (needs help) | 8.8
  Month 6: Cont (continent): number analyzed (Participants) | 259
  Month 6: Cont (continent) | 89.6
  Month 6: Cont (occasional incontinence): number analyzed (Participants) | 259
  Month 6: Cont (occasional incontinence) | 10.0
  Month 6: Cont (permanent incontinence): number analyzed (Participants) | 259
  Month 6: Cont (permanent incontinence) | 0.4
  Month 6: Feeding (self-sufficient): number analyzed (Participants) | 260
  Month 6: Feeding (self-sufficient) | 94.6
  Month 6: Feeding (needs help): number analyzed (Participants) | 260
  Month 6: Feeding (needs help) | 5.4
  Month 12: Bathing (self-sufficient): number analyzed (Participants) | 201
  Month 12: Bathing (self-sufficient) | 83.1
  Month 12: Bathing (partial help): number analyzed (Participants) | 201
  Month 12: Bathing (partial help) | 11.4
  Month 12: Bathing (washing impossible): number analyzed (Participants) | 201
  Month 12: Bathing (washing impossible) | 5.5
  Month 12: Dressing (self-sufficient): number analyzed (Participants) | 200
  Month 12: Dressing (self-sufficient) | 88
  Month 12: Dressing (partial help): number analyzed (Participants) | 200
  Month 12: Dressing (partial help) | 7.0
  Month 12: Dressing (completely undressed): number analyzed (Participants) | 200
  Month 12: Dressing (completely undressed) | 5.0
  Month 12: Toileting (self-sufficient): number analyzed (Participants) | 200
  Month 12: Toileting (self-sufficient) | 91.5
  Month 12: Toileting (needs help): number analyzed (Participants) | 200
  Month 12: Toileting (needs help) | 6.5
  Month 12: Toileting (doesn't go): number analyzed (Participants) | 200
  Month 12: Toileting (doesn't go) | 2.0
  Month 12: Transfer (self-sufficient): number analyzed (Participants) | 201
  Month 12: Transfer (self-sufficient) | 85.1
  Month 12: Transfer (needs help): number analyzed (Participants) | 201
  Month 12: Transfer (needs help) | 11.9
  Month 12: Transfer (bedridden): number analyzed (Participants) | 201
  Month 12: Transfer (bedridden) | 3.0
  Month 12: Cont (continent): number analyzed (Participants) | 197
  Month 12: Cont (continent) | 89.3
  Month 12: Cont (occasional incontinence): number analyzed (Participants) | 197
  Month 12: Cont (occasional incontinence) | 9.1
  Month 12: Cont (permanent incontinence): number analyzed (Participants) | 197
  Month 12: Cont (permanent incontinence) | 1.5
  Month 12: Feeding (self-sufficient): number analyzed (Participants) | 198
  Month 12: Feeding (self-sufficient) | 91.4
  Month 12: Feeding (needs help): number analyzed (Participants) | 198
  Month 12: Feeding (needs help) | 7.1
  Month 12: Feeding (complete help): number analyzed (Participants) | 198
  Month 12: Feeding (complete help) | 1.5
  Month 24: Bathing (self-sufficient): number analyzed (Participants) | 104
  Month 24: Bathing (self-sufficient) | 89.4
  Month 24: Bathing (partial help): number analyzed (Participants) | 104
  Month 24: Bathing (partial help) | 6.7
  Month 24: Bathing (washing impossible): number analyzed (Participants) | 104
  Month 24: Bathing (washing impossible) | 3.8
  Month 24: Dressing (self-sufficient): number analyzed (Participants) | 104
  Month 24: Dressing (self-sufficient) | 91.3
  Month 24: Dressing (partial help): number analyzed (Participants) | 104
  Month 24: Dressing (partial help) | 3.8
  Month 24: Dressing (completely undressed): number analyzed (Participants) | 104
  Month 24: Dressing (completely undressed) | 4.8
  Month 24: Toileting (self-sufficient): number analyzed (Participants) | 104
  Month 24: Toileting (self-sufficient) | 93.3
  Month 24: Toileting (needs help): number analyzed (Participants) | 104
  Month 24: Toileting (needs help) | 6.7
  Month 24: Transfer (self-sufficient): number analyzed (Participants) | 104
  Month 24: Transfer (self-sufficient) | 86.5
  Month 24: Transfer (needs help): number analyzed (Participants) | 104
  Month 24: Transfer (needs help) | 13.5
  Month 24: Cont (continent): number analyzed (Participants) | 104
  Month 24: Cont (continent) | 90.4
  Month 24: Cont (occasional incontinence): number analyzed (Participants) | 104
  Month 24: Cont (occasional incontinence) | 9.6
  Month 24: Feeding (self-sufficient): number analyzed (Participants) | 104
  Month 24: Feeding (self-sufficient) | 91.3
  Month 24: Feeding (needs help): number analyzed (Participants) | 104
  Month 24: Feeding (needs help) | 6.7
  Month 24: Feeding (complete help): number analyzed (Participants) | 104
  Month 24: Feeding (complete help) | 1.9

6. Secondary Outcome: Lawton Instrumental Activities of Daily Living Score (IADL)
Description: The Lawton Instrumental Activities of Daily Living Scale (IADL) is an appropriate instrument to assess independent living skills. The instrument is most useful for identifying how a participant is functioning at the present time and for identifying improvement or deterioration over time. There are 8 domains of function measured with the Lawton IADL scale (telephone use, shopping, cooking, housekeeping, laundry, mode of transportation, responsibility of own medications, and ability to handle finances). Participants are scored according to their level of functioning from 0 (low function, dependent) to 8 (high function, independent). Higher score for each domain represents better functional performance of the older people.
Time Frame: Baseline, Month 6, 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
units on a scale
  Baseline: number analyzed (Participants) | 343
  Baseline | 0.9 (1.1)
  Month 6: number analyzed (Participants) | 259
  Month 6 | 1.0 (1.2)
  Month 12: number analyzed (Participants) | 194
  Month 12 | 1.0 (1.2)
  Month 24: number analyzed (Participants) | 100
  Month 24 | 0.8 (1.2)

7. Secondary Outcome: Percentage of Participants With Balducci Score
Description: Balducci score defines an algorithm for the individual participant according to age, ADL and modified IADL 4-items scores, estimated performance status and comorbidities, particularly cardiovascular, cancer, depression or anemia. Balducci score is categorized in the following- Type 1 (Harmonious), Type 2 (Intermediate) and Type 3 (Frail). Type 1 indicates better results and Type 3 indicates worse outcomes.
Time Frame: Baseline, Month 6, 12, 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 358
Percentage of participants
  Baseline: Don't know: number analyzed (Participants) | 356
  Baseline: Don't know | 36.8
  Baseline: Type 1 (Harmonious): number analyzed (Participants) | 356
  Baseline: Type 1 (Harmonious) | 38.8
  Baseline: Type 2 (Intermediate): number analyzed (Participants) | 356
  Baseline: Type 2 (Intermediate) | 21.1
  Baseline: Type 3 (Frail): number analyzed (Participants) | 356
  Baseline: Type 3 (Frail) | 3.4
  Month 6: Don't know: number analyzed (Participants) | 260
  Month 6: Don't know | 37.3
  Month 6: Type 1 (Harmonious): number analyzed (Participants) | 260
  Month 6: Type 1 (Harmonious) | 36.9
  Month 6: Type 2 (Intermediate): number analyzed (Participants) | 260
  Month 6: Type 2 (Intermediate) | 22.3
  Month 6: Type 3 (Frail): number analyzed (Participants) | 260
  Month 6: Type 3 (Frail) | 3.5
  Month 12: Don't know: number analyzed (Participants) | 206
  Month 12: Don't know | 33.0
  Month 12: Type 1 (Harmonious): number analyzed (Participants) | 206
  Month 12: Type 1 (Harmonious) | 39.8
  Month 12: Type 2 (Intermediate): number analyzed (Participants) | 206
  Month 12: Type 2 (Intermediate) | 19.4
  Month 12: Type 3 (Frail): number analyzed (Participants) | 206
  Month 12: Type 3 (Frail) | 7.8
  Month 24: Don't know: number analyzed (Participants) | 99
  Month 24: Don't know | 27.3
  Month 24: Type 1 (Harmonious): number analyzed (Participants) | 99
  Month 24: Type 1 (Harmonious) | 50.5
  Month 24: Type 2 (Intermediate): number analyzed (Participants) | 99
  Month 24: Type 2 (Intermediate) | 16.2
  Month 24: Type 3 (Frail): number analyzed (Participants) | 99
  Month 24: Type 3 (Frail) | 6.1

ADVERSE EVENTS:
Time Frame: Up to 53 months
Description: Safety population included all participants who had at least one infusion of bevacizumab. The data in the study was collected for overall participants and not as per dose administered to participants.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 98/383
Other Adverse Events (participants affected / at risk) | 169/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=383)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Jugular Vein Thrombosis (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 2
Subclavian Vein Thrombosis (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Haematemesis (Gastrointestinal disorders) | 1
Ileal Fistula (Gastrointestinal disorders) | 1
Intestinal Ischaemia (Gastrointestinal disorders) | 1
Haemorrhagic Stroke (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 2
Leukoencephalopathy (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Acute Coronary Syndrome (Cardiac disorders) | 1
Anal Abscess (Infections and infestations) | 1
Anastomotic Fistula (Injury, poisoning and procedural complications) | 1
Haematuria (Renal and urinary disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Rectal Obstruction (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 2
Anal Fissure (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Gastrointestinal Toxicity (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Intestinal Perforation (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 4
Device Related Infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Ophthalmic Herpes Zoster (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonal Sepsis (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Subcutaneous Abscess (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
General Physical Health Deterioration (General disorders) | 11
Asthenia (General disorders) | 3
Death (General disorders) | 2
Face Oedema (General disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vena Cava Thrombosis (Vascular disorders) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3
Metabolic Alkalosis (Metabolism and nutrition disorders) | 1
Metabolic Disorder (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Renal Failure Acute (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Presyncope (Nervous system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Prothrombin Time Ratio Decreased (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional State (Psychiatric disorders) | 1
Psychiatric Symptom (Psychiatric disorders) | 1
Dihydropyrimidine Dehydrogenase Deficiency (Congenital, familial and genetic disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Hepatectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=383)
Anaemia (Blood and lymphatic system disorders) | 30
Neutropenia (Blood and lymphatic system disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 78
Nausea (Gastrointestinal disorders) | 37
Asthenia (General disorders) | 68
Vomiting (Gastrointestinal disorders) | 21
Fatigue (General disorders) | 21
Mucosal inflammation (General disorders) | 26
Decreased appetite (Metabolism and nutrition disorders) | 25
Neuropathy peripheral (Nervous system disorders) | 29
Hypertension (Vascular disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.